CLINICAL TRIAL: NCT02882776
Title: The Effect of Daily Ginger Drinking on Platelet's Function in the Saudi Population
Brief Title: Daily Ginger Drinking and Platelet Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC12/080
Record Dates: First submitted 2016-08-10; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Platelets Dysfunction; Hematological Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger drink once daily (Other): this group will receive ginger drink made by dissolving 4g ginger powder in plain water once a day for continuous 5 days.
  Interventions: Dietary Supplement: Ginger drink
- Ginger drink twice daily (Other): this group will receive ginger drink made by dissolving 4g ginger powder in plain water twice a day for continuous 5 days.
  Interventions: Dietary Supplement: Ginger drink

INTERVENTIONS:
Dietary Supplement: Ginger drink — Ginger powder dissolved in water

SUMMARY:
This study aims to examine the effect of ginger beverage consumption on platelets activity in apparently healthy Saudi adult volunteers.

As for the Saudi population, consumption of powdered ginger dissolved in hot water is a common practice. Accordingly, in this study, it is tempting to speculate the effect of this form of ginger consumption, given in separate time points per day, on platelet aggregation profile by using platelet aggregation analogues. If positive results were obtained, the herb could provide natural protection against the development of platelet aggregation complications and could be a potential alternative to aspirin, used for improving blood circulation and hematological pathophysiologies in diseased individuals.

DETAILED DESCRIPTION:
Herbal medicine products are dietary supplements that people take to improve their health. Many herbs have been used for a long time for claimed health benefits. They are sold as tablets, capsules, powders, beverages, extracts and fresh or dried plants. Herbal medicines have been associated with treatment of several physiological disorders of which hematological, mainly clotting disorders. Those include garlic, onion, and ginger in addition to pharmacological reagents such as aspirin, warfarin, heparin, and others. One of the herbal medications affecting hematological profile is ginger which has gained focus throughout studies conducted in previous years in the field of inhibiting platelet aggregation, taking benefit from some undesirable side effects arising from the use of other anti-platelet aggregation agents, especially aspirin.

Ginger (Zingiber officinale) is a well known spice and flavoring agent used in traditional medicine in many countries. It is a source of valuable phytonutrients characterized by having aromatic odor and pungent taste. The ginger rhizome contains 60% starch, 10%proteins, 10% fats, 5% fibers, 6% inorganic material, 10% residual moisture, 1-4% essential oils including gingerol and zingiberene, in addition to pungent principles such as zingerone, gingerol and shogaol. Shogaols are produced by heating gingerols. It has been speculated that ginger can eliminate symptoms associated with a variety of illnesses since there are a variety of chemical classes that these compounds belong to. Ginger has been used in the management of headache, nervous diseases, nausea, and vomiting. It has also been used to treat migraine headaches without side-effects. In addition, it is recommended in the management of rheumatic disorders and muscular pain. Ginger also acts as a metabolic enhancer where acetone extracts of ginger have stimulated bile secretion and excretion of gallstones. Although ginger is considered a safe herbal medicine with only few and insignificant adverse side effects, few undesirable effects like heartburn were noticed. In quantities higher than 6 g ginger may act as a gastric irritant and inhalation of dust from ginger may produce immunoglobulin E (IGE)-mediated allergy.

As for ginger toxicity, an acute overdose of ginger is usually in excess of about 2g of ginger per kilogram of body mass depending on the ginger tolerance level and can result in a state of central nervous system over-stimulation called "ginger gitters".

Experimental data reveals that ginger may be a dual inhibitor of eicosanoid synthesis, inhibiting the synthesis of both prostaglandins and leukotrienes, which are inflammatory mediators produced from arachidonic acid. With reference to the fact that normal platelet functioning is linked to an interplay between those substances, ginger consumption appears to be linked with reducing platelet aggregation.

Platelets have traditionally been linked with concepts of hemostasis and hemorrhagic disorders. However, with increasing incidence of atherosclerosis and hematologic disorders, the critical role played by platelets is more evident. Platelets are no longer viewed as "scaffolding" for the events of the coagulation cascade but rather as important catalysts in hemostasis, thrombosis, and fibrinolysis. Improved understanding of platelet physiology has led to developments of pharmacologic adjuncts resulting in improved patency rates and improved patient outcomes. Platelets are the smallest components in the blood stream, where they exist as a-nucleate disc-shaped cells in their resting state and travel singly as discoidal particles. In the presence of stimuli such as arachidonic acid, activated platelets change shape into spiny spheres. They bind to fibrinogen, aggregate and release the contents of their intracellular granules, including adenosine diphosphate (ADP) and serotonin.

ADP and an arachidonic acid (AA) metabolite acting an endogenous platelet activator, thromboxane A2 (TxA2), intensify the extent of platelet aggregation. ADP, arachidonic acid, epinephrine, and collagen act as agonists for platelet aggregation and clumping. These substances act in positive feedback loops, making platelet aggregation an autocatalytic rather than equilibrium response. Under pathophysiological conditions, platelet activation may result in peripheral, cardiovascular or cerebrovascular thrombosis with serious consequences.

Aspirin has been the main anti-platelet therapeutic agent. Inhibition of platelet aggregation by aspirin significantly reduces the incidence of first myocardial infarction, recurrent infarction and vascular death among patients with cardiovascular disease. Aspirin also reduces the risk of nonfatal stroke, nonfatal myocardial infarction and vascular death in patients with possible risk factors. However, aspirin ingestion, is mainly associated with gastric ulcers and gastrointestinal bleeding. Thus, the use of aspirin may be confined to elderly patients whose benefits outweigh increased risks of gastrointestinal bleeding.

Gingerols and their derivatives, especially [8]-paradol, have been reported to be more potent anti-platelet and cyclo-oxygenase-1 (COX-1) inhibitors than aspirin, when tested in vitro by the Chrono Log whole blood platelet aggregometer. Note that COX-1 is the enzyme responsible for the conversion of arachidonic acid into important biological mediators including prostaglandins, prostacyclins, and thromboxanes. These authors proposed that the carbonyl functional group at C3 found in paradol and in the diarylheptanoid series may contribute to their potent anti-platelet activity and inhibition of COX-1. Inhibition of the arachidonic acid (AA) metabolism cascade via the COX-1/thromboxane synthase system by these phenolic compounds may underline the mechanism of their action. In 2001 Koo et al. compared the ability of gingerols and related analogs to that of aspirin in inhibiting AA-induced human platelet serotonin release in vitro. Using the same dose range, it has been found that gingerols and related analogs were approximately two- to three-fold less potent than aspirin against the platelet release reaction initiated by AA, and two- to four-fold less potent than aspirin at inhibiting AA-induced platelet aggregation. Gingerols inhibited COX activity, assessed by measuring prostaglandin D2, a product of AA metabolism by COX. These results suggest that inhibition of COX activity by gingerols and related analogs may be the underlying mechanism for their effect on AA-induced platelet activation. 6-gingerol inhibits arachidonic acid-induced platelet aggregation and formation of thromboxane B2 and prostaglandin D2. Gingerol, shogaol and other structurally related substances in ginger inhibit prostaglandin and leukotriene biosynthesis.

Of the earlier studies conducted on ginger was that of Srivastava et al. in 1986 where they found that 5g of fresh, raw ginger has inhibited thromboxane B2 formation.

Furthermore, a study done on 20 healthy male individuals that were given 50 g of butter and 5g of ginger a day for seven days showed that addition of ginger with a fatty meal inhibited the platelet aggregation induced by adenosine diphosphate and epinephrine greatly. Ginger has been reported to inhibit prostaglandin synthesis in vitro. Dietary fat content affects platelet aggregation by modifying prostaglandin metabolism. Administration of ginger in a fatty diet inhibits the transformation of arachidonic acid to thromboxane and decreases the sensitivity of platelets to many aggregating agents. In 1994, Lumb et al., have shown in a cross over study conducted on 8 subjects that 2g of powdered ginger (prepared as medication) had no effect on bleeding time and whole blood platelet aggregation. Similarly, 15g and 40g of fresh or cooked raw ginger did not induce platelet aggregation in a cross over study conducted by Janssen et al. in 1996. Moreover, in 1997, Boardia et al. found that 4g of ginger powder was ineffective, where as 10g reduced platelet aggregation. Tested via addition of platelet aggregation agonists collagen, ADP, and epinephrine, platelet aggregation was inhibited by 35.3%, 37.8%, and 35.9% respectively upon administration of 1g dry ginger for a week. A combination of 1 g ginger with 10 mg nifedipine per day could be valuable for cardiovascular and cerebrovascular complication due to platelet aggregation.

Therefore, studies conducted to study the effect of ginger on bleeding risk have found no effect up to 15g raw ginger, 40g cooked ginger, or 4g dried ginger daily on platelet aggregation whereas 10g of dried ginger decreased platelet aggregation.

Throughout previous years, several studies have been designed to study the effect of different doses of different ginger forms (fresh, dry, extract, capsules) on platelet aggregation profile. Although most of them have made the suspect true, still others possess controversial results. In view of what literature has offered, it is most probable that ginger anti-platelet effect could be dose dependent, form dependent, and probably population or individual dependent as postulated by Helgason et al. in 1993 in their analysis of aspirin and warfarin platelet aggregation effect. Previous studies might have also employed old, non-reliable techniques in studying platelet aggregation profiles. As for the Saudi population, consumption of powdered ginger dissolved in hot water is a common practice. Accordingly, in this study, it is tempting to speculate the effect of this form of ginger consumption, given in separate time points per day, on platelet aggregation profile by using platelet aggregation analogues. If positive results were obtained, the herb could provide natural protection against the development of platelet aggregation complications and could be a potential alternative to aspirin, used for improving blood circulation and hematological pathophysiologies in diseased individuals.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy Saudi volunteers of either sex
* Age group = 18-60 years.

Exclusion Criteria:

* History of organ abnormalities or concomitant illnesses.
* Abnormal platelets count or function.
* Individuals with bleeding disorder as Von Willebrand Disorder or Hemophilia.
* Known allergy to ginger.
* Concurrent warfarin ingestion.
* History of ingestion of asprin,clopidogrel, nifedipine, non-steroid anti-inflammatory drugs (NSAIDs) or ethanol within the past two week.
* Any volunteer ingests ethanol, aspirin, clopidogrel, wine, beer and contraceptive pills during the study duration will be excluded from the study.
* pregnant & lactating women.
* Individuals on herbal treatment.
* Active G.I ulcers/ recently diagnosed G.I ulcers within one month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The effect of ginger beverage consumption on platelets activity will be examined in apparently healthy, Saudi adult volunteers. | 1 year

SECONDARY OUTCOMES:
The demographic characteristics of the sample under study will be identified. | 1 year
Any change in platelet morphology before and after ginger consumption will be studied | 1 year
Platelets' count before and after ginger consumption will be compared. | 1 year
Any change in platelets function after ginger consumption via addition of aggregation analogues will be studied. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Askar S. Alaskar, MD,FACP,FRCP, Principal Investigator — King Abdullah Medical research Center - King Abdulaziz Medical City - Riyadh
Locations (1):
- King Abdulaziz Medical City - National Guard Hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Undecided